CLINICAL TRIAL: NCT01492777
Title: Stabilization of Anticoagulation by Acenocoumarol: Role of Genetic Vulnerability and Risk of Drug Interactions
Brief Title: Pharmacogenetics of Acenocoumarol
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Jules Desmeules, Prof, University Hospital, Geneva
Other Study IDs: CER 08-019
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Thromboembolic Diseases

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The use of oral anticoagulation is marked by an elevated risk of adverse drug events (ADE) due to a narrow therapeutic window leading to important medical and economical consequences. The risk of ADE is increased partly by drug interactions and recently identified genetic factors influencing the metabolism of coumarins (polymorphism of the cytochrome P450 CYP2C9) as well as the target enzyme of the coumarins (polymorphism of the vitamin K epoxide reductase complex subunit 1 (VKORC1).

The objective is to determine the impact of several genotypes on acenocoumarol treatment and on vulnerability to drug-drug interactions.

ELIGIBILITY:
Inclusion Criteria:

* Every patients with requiring acenocoumarol therapy for at least 4 weeks and a target INR in the low intensity range (INR range 2-3)
* Age ≥ 18 years
* Signed informed consent

Exclusion Criteria:

* Severe cognitive impairment
* Previous or current treatment with any coumarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients starting acenocoumarol therapy
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2008-11; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Time to achieve stable dosing in days, since the beginning of the anticoagulation | 5 weeks

SECONDARY OUTCOMES:
Number of patients with INR > or = 4.0, which indicates overanticoagulation | 5 weeks
Time to achieve two consecutive therapeutic INRs | 5 weeks
Mean daily dosage of acenocoumarol | 5 weeks
Major bleedings and minor bleedings | 5 weeks
Thromboembolic events due to infratherapeutic anticoagulation | 5 weeks
Length of hospitalisation in days | 5 weeks
Potential of other drug interactions, linked to the observed genotype and phenotype of the patient | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jules A Desmeules, Prof, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospitals, Geneva, Switzerland

REFERENCES:
- [Derived] Gschwind L, Rollason V, Boehlen F, Rebsamen M, Combescure C, Matthey A, Bonnabry P, Dayer P, Desmeules JA. P-glycoprotein: a clue to vitamin K antagonist stabilization. Pharmacogenomics. 2015 Jan;16(2):129-36. doi: 10.2217/pgs.14.164. PMID 25616099